CLINICAL TRIAL: NCT02379260
Title: Development of a Therapeutic Education Intervention Improving Sexuality in Patients With Prostate Cancer Treated With Radical Prostatectomy
Brief Title: Development of a Therapeutic Education Program for Patients Operated for Prostate Cancer
Acronym: PEPs PROSTATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de la Loire (Other)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-11
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interview (Other): Patients and urologists will be interview by a sociologist.
  Interventions: Other: Interview with a sociologist
- Focus Groups (Other): Focus groups contain 5-7 patients. Groups will be stratified according to socio-economic levels and according to treatment (radical prostatectomy with conservation or without preservation of the neuro vascular strips).
  Interventions: Other: Interview with a sociologist

INTERVENTIONS:
Other: Interview with a sociologist

SUMMARY:
The aim is to built a Therapeutic Education Program for patients treated with radical prostatectomy in order to improve their sexuality.

This study is carried out in two steps :

* Identification of specific educational objectives through a sociological study, with interviews and focus groups conducted and analyzed by a sociologist. Patients from the urology department of the hospital center (CH) Lyon Sud - Hospices Civils de Lyon (HCL) will be included
* Development of the program by a caregiver education expert (Centre Hygée), adapted partly from results of the qualitative study and partly from concepts and tools from the Education Sciences.

DETAILED DESCRIPTION:
8 patients and 2 urologists will be interview to explore the educational needs and to create, expand and validate an interview guide. Exploratory interviews with urologists will address information given to patients on post radical prostatectomy sexual dysfunction, prescribing practices, monitoring therapy (PDE5 inhibitors, IIC, Vacuum), and patients adverse effects management.

Focus groups will be conduct to :

* Identify the representations associated with erectile dysfunction
* Identify the representations related to treatments for erectile dysfunction.
* Score patient knowledge about treatments and their managements.
* Identify common or original strategies to improve adherence, reduce side effects and overcome the disadvantages of the treatments.
* Assessing the needs and expectations of patients

ELIGIBILITY:
Inclusion Criteria:

* Patients followed in urology department Lyon Sud CH:
* Aged over 18 year
* Having a prostate cancer
* Treated with radical prostatectomy with or without conservation strips neuro vascular
* More than 1 month postoperative
* Having a normal preoperative erectile function defined by a score IIEF EF ≥ 26.
* And who signed the informed consent form for participation in the study

Exclusion Criteria:

* Score preoperative IIEF EF <26
* Refusal of participation, signed consent major patients protected under guardianship.
* Patients unable to understand the course of the study
* Patient (s) with a documented history of cognitive or psychiatric disorders.
* Geographical remoteness of more than 100 Kms.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Thematic and comparative analysis of the recorded interviews | 2 hours
  Thematic and comparative analysis of the recorded interviews and transcribed favoring a thematic approach that linked the different elements of speech.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Etienne TERRIER, MD, Principal Investigator — CH Lyon Sud
Locations (1):
- CH Lyon Sud, Pierre-Bénite, France